CLINICAL TRIAL: NCT02697318
Title: Evaluation of a New Method for Instilling Eye Drops
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Waterloo (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 21282
Record Dates: First submitted 2016-02-29; First posted 2016-03-03 (Estimated); Last update posted 2018-01-23 (Actual); Status verified 2018-01

CONDITIONS: Ophthalmic Solutions; Glaucoma
MeSH Terms: conditions — Glaucoma | interventions — Timolol; Ophthalmic Solutions

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Professional Administration (Other): Instillation of Timolol maleate 0.5% ophthalmic solution (or participant's own glaucoma medication) administered by a professional, using the standard clinical method.
  Interventions: Drug: Timolol maleate 0.5% ophthalmic solution
- Self-Administration (new method) (Other): Instillation of Timolol maleate 0.5% ophthalmic solution (or participant's own glaucoma medication) self-administered by the participant, using the new proposed method.
  Interventions: Drug: Timolol maleate 0.5% ophthalmic solution

INTERVENTIONS:
Drug: Timolol maleate 0.5% ophthalmic solution

SUMMARY:
The purpose of this project is to demonstrate that there is a new easier method to instill eye drops in ones own eye that is as effective as applying a drop directly to their open eye. The benefits of this new method include better medication compliance and reduced patient anxiety from instilling their eye drops. This secondary benefit should remove the "approach-avoidance response" that prompts some patients to delay or give-up on instilling their drops just to avoid the angst and frustration produced by the challenge.

The new method involves the patient instilling the eye drop onto their closed eyelid and then blinking the eye drop into their eye. We aim to show that this method has a similar therapeutic effect as the routine administration of an eye drop to an open eye.

DETAILED DESCRIPTION:
PURPOSE:

The purpose of this project is to test an alternative method for instilling eye drops. The new method involves the patient self-administer the eye drop onto the skin of their medial canthus, with the lids gently closed, and then open the lids once the "cold and wet" sensation of the eye drop is felt along the margins of the closed lids. We will compare the physiological and therapeutic efficacy of instilling the same eye drops into the eyes of the same subjects, using two methods. The first will be to have the eye drop administered using the "gold standard" method employed by optometrists to instill eye drops in the office. The second will be to employ the new method of self-administration described above.

HYPOTHESIS:

Instillation of an eye drop, over the gently closed lids at the medial canthus, has the same physiological effect and therapeutic efficacy as a drop of the same agent, at the same concentration, properly applied onto an open eye by a trained professional.

Aim #1: Determine if there is a difference in efficacy between drops of 0.5% timolol maleate administered by a professional, using the standard clinical method versus patient self-administration using the newly proposed method, in NORMAL SUBJECTS.

Aim #2: Determine if there is a difference in efficacy between glaucoma drops administered by a professional, using the standard method versus with patient self-administration of the same drop, using the newly proposed method, in GLAUCOMA PATIENTS.

JUSTIFICATION:

While new drug development in the glaucoma field seeks to address the issue of the difficulty patients experience with self-administration of an eye drop by pressing for new drugs that show efficacy in a once daily dosing routine, this strategy has potentially serious negative consequences. Clearly, when glaucoma medications are administered only once a day, if the patient misses their eye on that single instillation, the period of lapsed treatment is 24 hours or more. If their disease worsens, either due to non-compliance with their treatment regimen or inability to instill an eye drop, they will require more follow up visits, additional medications, additional diagnostic tests, and earlier surgery.

In this regard, the consequences of non-compliance or inability to comply are the same - increased blindness from glaucoma and increased costs associated with trying to prevent this blindness in needlessly advancing disease.

OBJECTIVES:

The objective of this proposal is to test the therapeutic efficacy of an alternative method of instilling eye drops. This requires comparing the effects of the same volume of the same drug, applied using the classical method and the new alternative method. If the proposed study is successful, a more reliable method for instilling drops of all kinds, to all patients, will have been validated.

ELIGIBILITY:
Aim #1:

Inclusion Criteria:

* both male and female participants are being studied
* minimum age of 21 and maximum age of 80
* healthy volunteers with no previous history of eye disease

Exclusion Criteria:

* no medical conditions representing contraindications to use of topical beta-blocker.
* subject must not have any active inflammatory diseases of the eye, or have a diagnosis of any form of glaucoma

Aim #2:

Inclusion Criteria:

* both male and female participants are being studied
* minimum age of 21 and maximum age of 80
* subjects have been diagnosed with primary open angle glaucoma and are stable on monotherapy

Exclusion Criteria:

- Subjects must have no other ocular disease, or a history of prior ocular trauma, beyond minor corneal abrasion or removal of a superficial corneal foreign body.

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-05; Primary Completion 2017-09 (Actual); Study Completion 2018-01-07 (Actual)

PRIMARY OUTCOMES:
Intraocular Pressure | 2 hours
  Intraocular Pressure by Goldmann applanation will be measured pre- and 2 hours post timolol maleate 0.5% ophthalmic solution

CONTACTS AND LOCATIONS:
Locations (1):
- University of Waterloo, Waterloo, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided